CLINICAL TRIAL: NCT05828277
Title: A Phase 1 Study to Assess the Effect of Hepatic Impairment on the Pharmacokinetics of Repotrectinib in Advanced Cancer Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Turning Point Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA127-1026; CA127-1026 (Other: BMS Protocol ID); TPX-0005-15 (Other: Turning Point Therapeutics Protocol ID)
Expanded Access: NCT05926232 (Available)
Record Dates: First submitted 2023-03-28; First posted 2023-04-25 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — repotrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Repotrectinib (TPX-0005) (Experimental): Oral repotrectinib (TPX-0005):
  Cohort 1: Patients with moderate hepatic impairment Cohort 2: Patients with severe hepatic impairment Cohort 3: Patients with normal hepatic function
  Interventions: Drug: repotrectinib (TPX-0005)

INTERVENTIONS:
Drug: repotrectinib (TPX-0005) — Oral repotrectinib (TPX-0005)
  Other Names: Oral TPX-0005 capsules; repotrectinib

SUMMARY:
This is a Phase 1 study to evaluate the effect of moderate or severe hepatic impairment on the PK of repotrectinib in patients with advanced cancer.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, multiple-dose, open-label, nonrandomized study to evaluate the effect of moderate or severe hepatic impairment on the PK of repotrectinib following single and multiple dose administration of repotrectinib in patients with advanced cancer. This study will enroll 8 patients each with moderate hepatic impairment, severe hepatic impairment and normal hepatic function.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumor for which standard curative or palliative measures do not exist or are no longer effective. In case of hepatocellular carcinoma, the diagnosis should be based on at least 1 of the following:

   1. The presence of at least 1 lesion, measuring ≥2 cm, with characteristic arterial enhancement and venous washout in the setting of liver cirrhosis and/or hepatitis B or C infection.
   2. The presence of liver lesion(s) (as defined in inclusion criteria 3a) with alphafetoprotein ≥ 400 ng/mL.
   3. Tissue confirmation.
2. For patients with genetic ROS1 or NTRK 1-3 gene fusion, tissue-based local testing should be documented.
3. Biliary obstruction for whom a biliary drain or stent has been placed are eligible.
4. Eastern Cooperative Oncology Group Performance Status scores 0 to 2.
5. The patient must have no clinically significant change in hepatic disease status within the last 30 days before screening.
6. Patient with ascites must not have a paracentesis within 3 months of screening.
7. Protocol specified baseline hematology and kidney function laboratory values

Key Exclusion Criteria:

1. Concurrent participation in another therapeutic clinical study.
2. Symptomatic brain metastases or leptomeningeal involvement.
3. Major surgery within 4 weeks.
4. Clinically significant cardiovascular disease.
5. History of non-pharmacologically induced prolonged QT interval corrected for heart rate interval.
6. Known active infections requiring ongoing treatment (bacterial, fungal, or viral, including human immunodeficiency virus positivity).
7. Gastrointestinal disease or other malabsorption syndromes.
8. Current use or anticipated need for drugs that are known to be strong cytochrome P450 (CYP) 3A inhibitors or inducers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) of repotrectinib | Within 22 days of first repotrectinib dose
  AUC0-t: Area under the plasma concentration-time curve from time 0 to the time of the last measurable concentration
Maximum Observed Plasma Concentration (Cmax) of repotrectinib | Within 22 days of first Repotrectinib dose
  Cmax: Evaluate the maximum plasma concentration

SECONDARY OUTCOMES:
Evaluate safety and tolerability | 28 days after last dose of repotrectinib
  To evaluate the safety and tolerability of repotrectinib in patients with moderate and severe hepatic impairment and patients with normal hepatic function following single and multiple dose administration of repotrectinib assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Gabrail Cancer Research Center, Canton, Ohio, United States
- Local Institution - 4103, Madrid, Spain